CLINICAL TRIAL: NCT02480322
Title: Metabolomic Fingerprint of Severe Obesity is Dynamically Affected by Bariatric Surgery in a Procedure-dependent Manner
Brief Title: Metabolomic Fingerprint After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: eSwiss Medical & Surgical Center (Other)
Collaborators: University of Florence (Other); FiorGen Foundation, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: Metab-001
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Obesity
Keywords: metabolic alterations
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- Sleeve group: Patients undergoing gastric sleeve resection.
  Interventions: Procedure: bariatric surgery (sleeve resection, proximal RYGB, distal RYGB)
- Proximal RYGB group: Patients undergoing proximal gastric bypass surgery.
  Interventions: Procedure: bariatric surgery (sleeve resection, proximal RYGB, distal RYGB)
- Distal RYGB group: Patients undergoing distal gastric bypass surgery.
  Interventions: Procedure: bariatric surgery (sleeve resection, proximal RYGB, distal RYGB)
- BMI-matched control group
- Normal-weight control group

INTERVENTIONS:
Procedure: bariatric surgery (sleeve resection, proximal RYGB, distal RYGB)
  Groups: Distal RYGB group; Proximal RYGB group; Sleeve group

SUMMARY:
Background: Obesity is associated with multiple diseases. Bariatric surgery is the most effective therapy for severe obesity that cannot only reduce body weight but also obesity-associated morbidity.

Objective: The metabolic alterations associated with obesity and respective changes after bariatric surgery are incompletely understood.

Design: In the longitudinal observational study, the investigator applied a 1H-NMR-based global, untargeted metabolomics strategy on human serum samples that were collected before and repeatedly up to one year after distinct bariatric procedures (sleeve gastrectomy, proximal and distal Roux-en Y gastric bypass; RYGB). For comparison, the investigator also analyzed serum samples from normal-weight and less obesity obese subjects that were matched for 1-year postoperative BMI values of the surgical groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/=35 kg/m2
* at least 2 years of unsuccessful conservative weight loss attempts

Exclusion Criteria:

* < 18 years of age
* BMI < 35 kg/m2
* informed consent was not signed by the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: severely obese patients of the Interdisciplinary Obesity Center, St. Gallen, Switzerland
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
compare the NMR metabolic fingerprint as assessed in serum samples of severely obese patients with that of normal-weight control subjects | pre operative
follow up changes in the metabolic fingerprint over one year after 3 distinct bariatric procedures | pre operative, 3-, 6-, 9- and 12 months post operative
compare the metabolic fingerprints established one year after the different surgeries with those of BMI-matched and normal-weight control subjects | 12 months post operative

REFERENCES:
- [Derived] Gralka E, Luchinat C, Tenori L, Ernst B, Thurnheer M, Schultes B. Metabolomic fingerprint of severe obesity is dynamically affected by bariatric surgery in a procedure-dependent manner. Am J Clin Nutr. 2015 Dec;102(6):1313-22. doi: 10.3945/ajcn.115.110536. Epub 2015 Nov 18. PMID 26581381